CLINICAL TRIAL: NCT02384525
Title: The Assessment of Volume Status by BIA and Lung Ultrasound in Septic AKI Patients Undergoing CRRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0791
Record Dates: First submitted 2015-02-26; First posted 2015-03-10 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Septic Acute Kidney Injury
Keywords: Septic AKI; CRRT; BIA
MeSH Terms: interventions — Electric Impedance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- clinical-based ultrafiltration (Experimental)
  Interventions: Procedure: Fluid management by the value of over hydration in Bioelectrical impedance
- BIA-based ultrafiltration (Active Comparator)
  Interventions: Procedure: Fluid management by clinical-based ultrafiltration

INTERVENTIONS:
Procedure: Fluid management by the value of over hydration in Bioelectrical impedance — In this study, investigator measure the fluid status of the patients by bioelectrical impedance analysis and lung ultrasound. The patients are assigned into two groups, BIA and Lung Ultrasound based versus clinical-based assessment group. Ultrafiltration of BIA and Lung Ultrasound based group is adjusted to be equal to the value of over hydration measured only by BIA, not by Lung Ultrasound, because Lung Ultrasound cannot determine exact amount of the patient's fluid excess. Total amount of ultrafiltration will be removed from the patient for three days evenly. On the other hand, Ultrafiltration amount will be decided by the physician in the clinical based group. Amount of fluid removal for a day will be adjusted not to exceed 2000ml, so that total fluid removed from the patient will not exceed 6000ml for three days.
  Arms: clinical-based ultrafiltration
Procedure: Fluid management by clinical-based ultrafiltration — In this study, investigator measure the fluid status of the patients by bioelectrical impedance analysis and lung ultrasound. The patients are assigned into two groups, BIA and Lung Ultrasound based versus clinical-based assessment group. Ultrafiltration of BIA and Lung Ultrasound based group is adjusted to be equal to the value of over hydration measured only by BIA, not by Lung Ultrasound, because Lung Ultrasound cannot determine exact amount of the patient's fluid excess. Total amount of ultrafiltration will be removed from the patient for three days evenly. On the other hand, Ultrafiltration amount will be decided by the physician in the clinical based group. Amount of fluid removal for a day will be adjusted not to exceed 2000ml, so that total fluid removed from the patient will not exceed 6000ml for three days.
  Arms: BIA-based ultrafiltration

SUMMARY:
Acute kidney injury(AKI) is one of the most common complications that occur up to 35% of critically ill patients. Septic AKI accounts for one third of them. Patients with septic AKI are widely treated with Continuous renal replacement therapy (CRRT). However, previous studies have hardly documented improvement of mortality in septic AKI patients. Otherwise, Fluid overload in septic shock patients who are undergoing CRRT is proven to be a significant predictor for mortality. Recent studies showed efficacy of bioelectrical impedance analysis and lung ultrasound in assessing fluid status of the patients. Thus, hypothesis of the study is that fluid assessment and control of fluid status using BIA and Lung Ultrasound could be related to the outcome of septic AKI patients who undergo CRRT. In this study, the investigators measure the fluid status of the patients by bioelectrical impedance analysis and lung ultrasound for experimental group, while for control group, fluid status would be determined clinically by the physician. Ultrafiltration rate of experimental group is adjusted to be equal to the value of overhydration measured by BIA.

ELIGIBILITY:
Inclusion Criteria:

1. body temperature < 36 °C or > 38 °C
2. heart rate > 90 BPM
3. respiratory rate > 20 or aPaCO2 < 32 mmHg on ABG
4. White blood cell count < 4,000 cells/mm3 or > 12,000 cells/mm3 or band forms (immature white blood cells) ≥10%
5. Evidence of infection
6. WBCs in normally sterile fluid
7. Perforated viscus
8. radiologically proven infection
9. more than Injury stage in AKI according to RIFLE criteria
10. septic AKI which is not explained by other cause
11. patients signed a written informed consent.

Exclusion Criteria:

1. Younger than 19 years old, older than 80 years old
2. Previously undergoing dialysis treatment due to ESRD
3. Underlying malignancy, Life expectancy shorter than 3 month
4. AKI due to other than sepsis
5. patients with intracardiac device such as Pacemaker, CRT, ICD

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
28-day all cause mortality | 28th day from CRRT

SECONDARY OUTCOMES:
Dialysis free rate | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea